CLINICAL TRIAL: NCT05607966
Title: A Post-market Observational ORIGIN® CR Clinical Study
Status: Recruiting | Type: Observational
Sponsor: Symbios Orthopedie SA (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-G-014
Record Dates: First submitted 2022-10-27; First posted 2022-11-07 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Total Knee Replacement
Keywords: ORIGIN; TKA; Prosthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ORIGIN® CR devices — It is planned to include consecutive eligible subjects which will be treated with the ORIGIN® CR devices.

SUMMARY:
The study objective is to evaluate safety and performance of the ORIGIN® CR (cruciate retaining) devices and associated instruments, more precisely to evaluate safety by the proportion of patients requiring a revision (i.e. revision rate) at 1-year post procedure and to evaluate performance by means of a Knee Society Score (KSS) Knee Score at 1 year post procedure and by means of a KSS Function Score also at 1 year post procedure.

The hypothesis raised for this study, regarding the scoring, is that patients will experience a marked improvement in the natural feel of the prosthesis during the first year after the surgery, and slightly significant improvement at the following interval of 2 years. The overall patient satisfaction is expected to be improved after 2 years follow-up with ORIGIN® CR.

DETAILED DESCRIPTION:
The study is a prospective, non-comparative, non-randomized, single-arm, observational, post market study in which 199 patients will be enrolled to evaluate the safety and performance of the ORIGIN® CR devices and associated instruments.

Patients will be included in the study during 18 months (inclusion window) and followed-up for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Male and female over 18 years of age
* Each patient who is willing to give informed consent.
* Clinically indicated for a total knee replacement
* Females who are not pregnant and not planning to become pregnant ≤ 12 months. A pregnancy test should be performed for women of childbearing age
* Geographically stable and willing to return to the implanting site for all follow-up visits at 1 year and 2 years.

Exclusion Criteria:

* Acute or chronic, local or systemic infection
* Muscular, ligamental, neurological, psychological or vascular deficits
* Bone destruction or poor bone quality likely to affect implant stability (requiring a femoral and/or a tibial stem and/or a thick insert)
* Any concomitant condition likely to affect implant integration or function
* Allergy or hypersensitivity to any of the materials used
* For devices in CoCrMo (ISO 5832/4): renal and hepatic impairment
* Hip Knee Ankle (HKA) angle < 165° or > 195°
* Severe collateral ligaments deficiency (requiring a more constrained prosthesis)
* Posterior cruciate ligament deficiency
* Major anatomical deformities
* Severe flexion contracture or severe recurvatum
* Revision of a partial or total knee prosthesis
* Non-extractible material (e.g. screws, plate, intramedullary nail, osteosynthesis material…) which can create a conflict with any component of the prosthesis
* Distal and/or posterior and/or anterior femoral bone loss which exceeds the femoral component thickness
* Proximal tibial bone loss which exceeds the tibial component thickness (tibial tray + tibial insert)
* Bone degradation requiring an anchoring stem for femoral component

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have provided consent for the collection of their data and met the protocol eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety by the proportion of required revisions | 1 year post-procedure
  Proportion of patients requiring a revision after 1-year post-procedure. The revision rate is consistent with the state of the art - Orthopaedic Data Evaluation Panel (ODEP) benchmark system (revision rate not higher than 2.5% to 3.5% at 1 year, 4% to 6% at 5 years and 5% to 7% at 10 years).
Evaluate performance | 1 year post-procedure
  Evaluate performance by means of following questionnaires: Knee Society Score (KSS) and a Knee Society Function score, a partient-reported outcome measure.
  The KSS contains questions in 2 sections: knee joint (pain, range of motion, stability) and function (walking distance, ability to climb stairs). When calculating the score, deductions are taken for assistive devices and flexion contractures, misalignment, or extension lag. The maximum points which can be reached are 100 points.
  * Clinical status assessed by means of the KSS Knee score at 1 year post procedure
  * Clinical status assessed by means of the KSS Function score at 1 year post procedure

SECONDARY OUTCOMES:
Evaluate safety by the proportion of required revisions | 2 years post procedure
  Proportion of patients requiring a revision after 2 years post-procedure.
Performance on patient satisfaction | 1- and 2-years post-procedure
  Patient satisfaction questionnaires at 1 year and 2 years follow-up visits.
Quality of Life post-procedure measured by the Knee Society score and Knee Society function questionnaire | 1- and 2-years post-procedure
  Quality of Life measured by means of the Knee Society score and Knee Society function score questionnaires at 1- and 2-years follow-up visit.
Quality of Life post-procedure measured by the Forgotten Joint Score questionnaire | 1- and 2- years post-procedure
  Quality of Life measured by means of the Forgotten Joint Score questionnaire at 1- and 2-years follow-up visit.
  12 questions refer to how aware the patients are of their artificial hip/knee joint in everyday life
  Scoring: For scoring the FJS-12, all responses are summed (never, 0 points; almost never, 1 point; seldom, 2 points; sometimes, 3 points; mostly, 4 points) and then divided by the number of completed items. This mean value is subsequently multiplied by 25 to obtain a total score range of 0 to 100.
  Finally, the score is subtracted from 100, to change the direction of the final score in a way that high scores indicate a high degree of "forgetting" the artificial joint, that is, a low degree of awareness.
  If more than 4 responses are missing, the total score should not be used.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - GZA Ziekenhuizen - campus Sint-Augustinus, Antwerp
  - AZ Voorkempen, Malle

IPD SHARING:
Plan to Share IPD: No